CLINICAL TRIAL: NCT00010387
Title: Phase II Study of High-Dose Cyclophosphamide in Patients With Severe Autoimmune Hematologic Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 199/15672; JHOC-J9881; JHOC-99012906
Record Dates: First submitted 2001-02-02; First posted 2001-02-02 (Estimated); Last update posted 2008-09-10 (Estimated); Status verified 2008-09

CONDITIONS: Anemia, Hemolytic, Autoimmune; Felty Syndrome; Purpura, Thrombocytopenic; Autoimmune Diseases
Keywords: Felty syndrome; autoimmune hemolytic anemia; autoimmune neutropenia; hematologic disorders; immune thrombocytopenic purpura; rare disease
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Felty Syndrome; Purpura, Thrombocytopenic; Autoimmune Diseases; Hematologic Diseases; Purpura, Thrombocytopenic, Idiopathic; Rare Diseases | interventions — Cyclophosphamide; Filgrastim

INTERVENTIONS:
Drug: cyclophosphamide
Drug: filgrastim

SUMMARY:
OBJECTIVES:

I. Determine the response rate and 1-year event-free survival in patients with severe autoimmune hematologic disease treated with high-dose cyclophosphamide.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Patients receive high-dose cyclophosphamide IV on days 1-4 and filgrastim (G-CSF) starting on day 10 and continuing until blood counts recover.

Patients are followed at 1, 3, 6, and 12 months and then annually thereafter.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of severe autoimmune hematologic disease Autoimmune hemolytic anemia OR Immune thrombocytopenia
* Failure of at least 2 standard treatment approaches (e.g., prednisone therapy, splenectomy, intravenous immunoglobulin, or other immunosuppressants)
* Inability to taper prednisone dose to less than 10 mg/day OR Autoimmune neutropenia including the following: Felty's syndrome OR Disorders of large granular lymphocytes with recurrent infections or absolute neutrophil count less than 200/mm3

--Prior/Concurrent Therapy--

* See Disease Characteristics

--Patient Characteristics--

* Age: Not specified
* Performance status: Not specified
* Hematopoietic: See Disease Characteristics
* Hepatic: Not specified
* Renal: Creatinine no greater than 2.5 mg/dL
* Cardiovascular: Ejection fraction at least 40%
* Pulmonary: FVC, FEV1, or DLCO at least 50% predicted

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Not preterminal or moribund

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32
Dates: Start 1999-03; Primary Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Brodsky, Study Chair — Johns Hopkins University
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States